CLINICAL TRIAL: NCT00552201
Title: Randomized Therapeutic Study of a Treatment by Tacrolimus Adapted or Not According to the Genotype of the Cytochrome P450 3A5 After Renal Transplantation
Brief Title: TACrolimus in Renal Transplantation: Individualization by Pharmacogenetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Roche Pharma AG (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIQUE
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; Tacrolimus; P450 3A5 cytochrome; genotype
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tacrolimus — Administration Twice a day after adjustment to blood level

SUMMARY:
Renal transplantation is the treatment of choice of the chronic renal insufficiency arrived at its final stage. Tacrolimus is an immunosuppressant treatment used for the prevention of episodes of acute rejection. Tacrolimus is characterized by a narrow therapeutic index and important interindividual variations of its pharmacokinetic characteristics. Proteins CYP3A4 and CYP3A5 are responsible of intestinal and hepatic metabolism of Tacrolimus. Various polymorphisms for CYP3A5 and CYP3A4 were described and several retrospective studies suggested an association between a genetic polymorphism of CYP3A5 and the pharmacokinetic parameters of Tacrolimus. In particular, we showed that the presence of an allele CYP3A5*1 was associated to the use of more important amounts of Tacrolimus to obtain the desired blood concentrations.

This study is a national, multicentric, prospective, opened, randomized on two arms of treatment. 280 receivers of a renal transplant in 12 centres will be included. The genotyping of gene CYP3A5 will be carried out in the 6 days following transplantation. During the first week, the patients will be treated by basiliximab, MMF and corticosteroids. They will be randomized (central randomization) in D6 to receive either Tacrolimus at 0.2 mg/kg/d, or at a dosage adapted to their genotype. After determination of the first residual blood concentration of Tacrolimus realized after six oral intakes, the daily amounts of Tacrolimus could be modified if necessary to reach the desired blood concentrations. The total duration of the study for a patient is 3 months after transplantation.

The objective of this study is to evaluate the impact of the adaptation, according to the genotype of the CYP3A5 of the patient, of the first amount of Tacrolimus on the first residual blood concentration of Tacrolimus, keeping in mind the aim of the individualization of dosage schedule by pharmacogenetic approach.

Principal criterion : Comparison, between the two groups, of the percentage of patients for whom the first blood concentration of Tacrolimus evaluated 3 days (D10) after the first administration of Tacrolimus ranges between 10 and 15 ng/ml.

Statistics will be carried out in intention to treat. The principal criterion will be analyzed by the test of chi-2.

DETAILED DESCRIPTION:
Inclusion criteria

* Patients, male or female, 18 to 65 years old.
* Patients receiving a first or a second isolated renal graft coming from a donor alive or deceased,
* The patients in age to procreate must have a negative test of pregnancy before being included in this study and will have to agree to use effective contraceptive measurements throughout the study.
* Patients able to include/understand the aims and the risks of the study, having been fully informed and having given their writing consent to take part in this study. Patients unable to write and/or read but having fully understood the oral information given by the investigator and having given their oral consent in the presence of an independent witness.

Non-inclusion criteria

* Patients who receive several grafts.
* Patients requiring a treatment by azathioprin.
* Pregnant woman or nursing mother
* Patients receiving an incompatible graft ABO.
* Patients receiving or requiring immunosuppressant drugs prohibited by the protocol.
* Patients with a peak of historical antibody equal to or greater than 50% of the panel.
* Patients suffering from serious gastro-intestinal disorders which interfere with their capacity to receive or to absorb an oral form and patients presenting severe diarrhoea.
* Patients with symptomatic GI ulcer
* HIV or HTLV1 positive patients or their donors
* Patients presenting or having presented in the 5 last years one or several malignant tumours, except baso or spinocellular cutaneous epithelioma successfully treated.
* Patients with systemic infections requiring a treatment at the entry in the study.
* Patients having a leukocyte numeration lower than 2,5.109/l or haemoglobin lower than 5g/dl.
* Patients with drug-addiction whatever it is, or psychiatric disorder which, according to the point of view of the investigator, could invalidate the communication with investigator or interfere with the compliance of the patient.
* Patients who take part simultaneously in another therapeutic test or who received a study treatment less than 30 days before the entry in this study.
* Patients having already been included in this study.
* Patients allergic or intolerant with corticoids, macrolides, Tacrolimus, mycophenolate mofetil or basiliximab

The inclusion period is planned for 15 month. The inclusion of the patients will take place before transplantation. After transplantation, a centralized genotyping of CYP3A5 will be carried out for each patient. A sample of blood will be taken the day of transplantation.

The randomization will be carried out according to a 1:1 mode, by unequal blocks and stratified on the center according to group A (Tacrolimus given at D7,dosage:0,20 mg/kg/d) versus group B (managed Tacrolimus given at D7 dosage adapted to genotype CYP3A).

VISITS

The participation of the patient in this study will be 3 months. For this period, 7 visits are planned. D0 being considered as the day of the closing of the skin.

* Before transplantation Visit 1: inclusion visit(in the 4 days before transplantation) The day of transplantation a blood taking will be carried out on EDTA tube for CYP 3 A5 genotyping
* After transplantation (D0 = day of closing of the skin)

  * Visit 2: J6 (randomization)
  * Visit 3: J10
  * Visit 4: J14
  * Visit 5: M1 + - 3 days
  * Visit 6: M2 + - 3 days
  * Visit 7: M3 + - 7 days

TREATMENTS:

-Tacrolimus In the two arms of treatment Tacrolimus will be given at D7 post transplantation according to the group of randomization.

The first dosage schedule of Tacrolimus will be different according to the group of randomization:

* Group A: 0,10 mg/kg 2 times per day for all the patients
* Group B:

  * 0,125 mg/kg 2 times per day (CYP3A5 *1/*1 or *1/*3)
  * 0,075 mg/kg 2 times per day (CYP3A5*3/*3)

A first residual blood concentration (C0) of Tacrolimus will be evaluated after 6 administrations of Prograf®, at D10. The dosage schedule of Tacrolimus will then be adapted freely according to the therapeutic pharmacological follow-up of Tacrolimus specified in the protocol, that is to say 10 to 15 ng/ml, whatever the group of randomization.

* Basiliximab All the patients will receive two injections of basiliximab per intravenous way (first injection before transplantation and second injection at D4),20 Mg by intake.
* Corticotherapy in decreasing amount as follows:

  * D0: 500 Mg
  * D1: 125 Mg
  * D2 - D15: 20 Mg
  * D16 - M1: 15 Mg
  * M1 - M3: 10 Mg
* MMF The MMF will be given 3 gr. per day during the first 15 days, then 2 G per day adapted according to the clinical and biological tolerance.

During this study the following treatments will not be authorized :

* immunosuppressants other than those proposed; ciclosporin, sirolimus, azathioprine, plasmatic exchanges; intravenous immunoglobulins.
* Gastric bandages [gastric protections (inhibitors of the H+ pump) are authorized].
* Treatments presenting an interaction with P-glycoprotein or cytochromes P450 3A
* Any drug not having a marketing authorization. All the concomitant drugs taken by the patient during this study must be written in the CRF as all the drugs the patient would have taken in the 7 days before transplantation.

The analysis of this test will be done at the end of the inclusion on all the patients according to the principle of Intention To Treat Analysis.

The patients being able to be excluded from this analysis will be:

* patients not having taken no amount of the evaluated drug
* patients without data collected after the randomization

An analysis per-protocol will be carried out. From this analysis could be excluded in an additional way to the preceding analysis:

* declared patients not compliants
* patients who left the study for another reason that the inefficiency of the treatment or an undesirable event
* patients having taken during the study one or more prohibited treatments which can influence the effectiveness.

STATISTIC

Calculation of the necessary number of subjects:

One defines as a success: The event "blood concentration of Tacrolimus is between 10 and 15 ng/ml after 6 administrations per bone" One defines as a failure: The event "blood concentration of Tacrolimus is not between 10 and 15 ng/ml after 6 administrations per bone".

The awaited percentage of event is 40% in group A (dosage schedule of Tacrolimus according to recommendations: 0,20/kg/d).

It is made the assumption that the adaptation of the dosage schedule of Tacrolimus according to genetics will increase the success rate to 60%.

By setting an alpha risk = 5%, a beta risk = 10%, in bilateral formulation, by balancing the randomization (1/1), it are necessary to include 140 subjects by group to show an absolute difference of 20% of success between the 2 groups, that is to say 1 year of inclusion and 1 year and 3 months of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, 18 to 65 years old.
* Patients receiving a first or a second isolated renal graft coming from a donor alive or deceased,
* The patients in age to procreate must have a negative test of pregnancy before being included in this study and will have to agree to use effective contraceptive measurements throughout the study.

-Patients able to include/understand the aims and the risks of the study, -having been fully informed and having given their writing consent to take part in this study. Patients unable to write and/or read but having fully understood the oral information given by the investigator and having given their oral consent in the presence of an independent witness. -

Exclusion Criteria:

* Patients who receive several grafts.
* Patients requiring a treatment by azathioprin.
* Pregnant woman or nursing mother
* Patients receiving an incompatible graft ABO.
* Patients receiving or requiring immunosuppressant drugs prohibited by the protocol.
* Patients with a peak of historical antibody equal to or greater than 50% of the panel.
* Patients suffering from serious gastro-intestinal disorders which interfere with their capacity to receive or to absorb an oral form and patients presenting severe diarrhoea.
* Patients with symptomatic GI ulcer HIV or HTLV1 positive patients or their donors
* Patients presenting or having presented in the 5 last years one or several malignant tumours, except baso or spinocellular cutaneous epithelioma successfully treated.
* Patients with systemic infections requiring a treatment at the entry in the study.
* Patients having a leukocyte numeration lower than 2,5.109/l or haemoglobin lower than 5g/dl.
* Patients with drug-addiction whatever it is, or psychiatric disorder which, according to the point of view of the investigator, could invalidate the communication with investigator or interfere with the compliance of the patient.
* Patients who take part simultaneously in another therapeutic test or who received a study treatment less than 30 days before the entry in this study.
* Patients having already been included in this study.
* Patients allergic or intolerant with corticoids, macrolides, Tacrolimus, mycophenolate mofetil or basiliximab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

SECONDARY OUTCOMES:
Severity of the delayed restart of the renal function evaluated by the number | 3 months
of dialysis; | 3 months
C0 of Tacrolimus at D14, M1, M2 and M3; | 3 months
AUC (0-12h) of Tacrolimus at D14, M1 and M3; | 3 months
Time (in D) to obtain C0 targets of Tacrolimus between 10 and 15 ng/ml | 3 months
Number of dosage schedule adjustments for Tacrolimus necessary to obtaining | 3 months
first C0 target between 10 and 15 ng/ml; | 1 month
Global frequency of the clinical acute rejections; | 3 months
Time and incidence of the first episode of acute rejection proven and not by biopsy | 3 months
Renal graft function at M1 and M3 evaluated by the calculated | 3 months
creatinin clearance; | 3 months
Survival of the patients at M3; | 3 months
Survival of the grafts at M3; | 3 months
Number of adverse events at M3; | 3 months
Pharmacoeconomic impact at M3 evaluated by the duration of the initial | 3 months
hospitalization, the need of care (dialysis, rejection acute, opportunist infection) the frequency and duration of the hospitalizations during the first 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Choukroun, MD, PhD, Principal Investigator — CHU Amiens; Eric Thervet, Md, PhD, Principal Investigator — Hôpital Necker, Paris
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHU Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - CHU de la côté de Nacre, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - CHU Poitiers- hôpital Jean Bernard, Poitiers
  - CHU Reims - Hôpital Maison Blanche, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Strasbourg - Hospices Civils, Strasbourg
  - CHU Tours - Hôpital Bretonneau, Tours

REFERENCES:
- [Background] Pallet N, Etienne I, Buchler M, Bailly E, Hurault de Ligny B, Choukroun G, Colosio C, Thierry A, Vigneau C, Moulin B, Le Meur Y, Heng AE, Legendre C, Beaune P, Loriot MA, Thervet E. Long-Term Clinical Impact of Adaptation of Initial Tacrolimus Dosing to CYP3A5 Genotype. Am J Transplant. 2016 Sep;16(9):2670-5. doi: 10.1111/ajt.13788. Epub 2016 Apr 8. PMID 26990694